CLINICAL TRIAL: NCT01909583
Title: Pediatric Cardiac Surgery Pre-operative Counselling Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. David Horne, Doctor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H2013:117
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Heart Disease
Keywords: congenital; surgery; peri-operative; counselling
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAGES PRE-GROUP (Active Comparator): INTERVENTION: this group will receive our "STAGES" booklet PRE-operatively
  Interventions: Other: STAGES-Booklet
- STAGES POST-GROUP (Placebo Comparator): INTERVENTION: This arm will only receive the STAGES-booklet POST-operatively
  Interventions: Other: STAGES-Booklet

INTERVENTIONS:
Other: STAGES-Booklet — STAGES-booklet was designed by the investigators focussing on guiding parents through the pre-operative and operative admission period.

SUMMARY:
We have developed a pre-operative educational / counselling booklet with the focus on informing parents / patients about the different stages before, during, and after cardiac surgery that they will encounter; both chronologically and emotionally. With this approach and study our objectives are:

1. To provide anticipatory guidance for parents to decrease parental stress and improve parental experience and preparedness, thus involving the parent as a partner in caring for their child.

We hypothesize that this additional tool will improve parental satisfaction in regards to being prepared for their child's heart surgery.

DETAILED DESCRIPTION:
Our study objectives are to provide anticipatory guidance for parents to decrease parental stress and improve parental experience and preparedness, thus involving the parent as a partner in caring for their child.

A Case-control trial comparing family satisfaction between families that did and did not receive the STAGES-booklet.

Primary endpoints are Family satisfaction score and Family stress score. Secondary endpoints are Percentage of families that would recommend the STAGES-booklet as routine pre-operative educational tool, as well as Family Stress score during each stage as outlined in the STAGES-booklet

The Study period either 1 year or once 100 participants enrolled have completed their post-operative survey

Methods Group allocation: The first 50 families will be assigned to the STAGES-post group, and the last 50 to the STAGES-pre group. In both groups participants will be blinded to their timing of exposure to the intervention. This randomization in an attempt to minimize educator bias of possibly giving the STAGES-post group information pertaining to the intervention proposed.

Time points: Routinely after the cardiologist informs families that their child has a cardiac condition needing intervention, the Variety Children's Heart Centre clinical resource nurses, meet with families to help them navigate through upcoming events, do pre-operative counselling and supply them with educational material. At this point parents will be asked in a sensitive manner, whether they would consent to taking part in this study (see consent form). The first 50 will be informed that they will receive a booklet (not disclosing the STAGES-booklet) post-operatively to evaluate and a survey to complete post-operatively. The subsequent 50 families will be given the STAGES-booklet (not disclosing that STAGES is the interventional tool being investigated) together with the other routine educational material, and be counselled according to the STAGES-philosophy. Before leaving the province for cardiac surgery, the RN's will in addition to logistical matters, repeat the STAGES-booklet review and teaching with the STAGES-pre group.During the routine post-operative visit at 6-12 weeks, families will be warned that their visit will be approximately 20-30 minutes longer to complete the post-operative evaluation-survey. The STAGES-post group will be given the STAGES-booklet and informed of the STAGES-philosophy before completing the post-operative survey.In both groups, parents will receive condition specific teaching that is part of routine care currently.

Data collection : Surveys will contain only the family's study number in order to remain anonymous. Data will be analyzed collectively at the end of the study.

Survey responses will be aggregated and appropriate statistical analysis performed by the CHARM statistician.

Expected outcomes:Mean Family satisfaction scores will be 10-20% higher, and mean emotional stress scores 10-20% lower in the STAGES-pre group compared to the STAGES-post group. More than 80% of families in each group will recommend the STAGES-booklet and/or philosophy to be used as a routine pre-operative tool.

Results will be published in a respectable influential journal, submitted to national and international conferences, with the goal to promote the use of STAGES, across Canada and internationally.

ELIGIBILITY:
Inclusion Criteria:

1. All consented families of children <18 years that will be sent out of province for cardiac surgery from the Variety Children's Heart Centre

Exclusion Criteria:

1. Families that can't read or write english

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Family satisfaction and stress score | up to 6 weeks post-operatively
  At post-operative visit families will complete a study questionnaire evaluating their satisfaction of pre-operative preparation and their stress levels during the surgical period

SECONDARY OUTCOMES:
Percentage of families that would recommend the STAGES-booklet as routine pre-operative educational tool. | 1 day (At post-operative visit)
Family Stress score during each stage as outlined in the STAGES-booklet | 1 day (At post-operative visit)

CONTACTS AND LOCATIONS:
Overall Officials: David Horne, MD, Principal Investigator — University of Manitoba
Locations (1):
- Variety Children's Heart Centre, Winnipeg, Manitoba, Canada